CLINICAL TRIAL: NCT00006146
Title: Evaluation of the Immunogenicity of Low Dose Trivalent Inactivated Influenza Vaccine in Healthy Adults
Brief Title: Half-Dose Flu Vaccine Study in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Prevention
Other Study IDs: DMID 00-009
Record Dates: First submitted 2000-08-07; First posted 2001-08-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Approved influenza virus vaccine.

SUMMARY:
It appears likely that there will be a delay and possibly a reduction in the amount of influenza vaccine available for the 2000-2001 influenza season. One possible way of increasing the availability of influenza vaccine for this year is to use a half-dose in healthy adults. The objective of this study is to determine if the immune system responds to a half-dose the same way it responds to a whole dose. This study will use the currently approved inactivated influenza vaccine in healthy adults ages 18 to 49 years old.

If the immune response to the half-dose is not significantly different than the immune response generated to the whole dose, this could be a strategy to extend the amount of vaccine that could be available in this age group.

DETAILED DESCRIPTION:
Eligible subjects will be randomized to receive a single intramuscular injection of either a half-dose or a whole dose of a currently approved influenza virus vaccine in their arm. Prior to vaccination, subjects will have one tube of blood drawn. Subjects will be given a 3-day diary card to record any symptoms they may experience and asked to return for a second and final visit approximately 21 days following vaccination. A second blood draw will be done.

ELIGIBILITY:
Inclusion Criteria:

Volunteers may be eligible for this trial if they:

* Are able to and have given informed consent.
* Are able to understand and comply with all study procedures and to complete study diary.
* Are aged 18 to 49 years.
* Are female, and are not pregnant.
* Are available for all study visits.

Exclusion Criteria:

Volunteers will not be eligible for this trial if they:

* Are allergic to eggs or egg products.
* Have a current chronic medical condition for which influenza vaccine is normally recommended.
* Have received experimental vaccines or medications within 30 days of study entry.
* Have received parenteral immunoglobulin within 30 days of study entry.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 840
Dates: Start 2000-08; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, Principal Investigator — Univ of Rochester Medical Center
Locations (6):
- United States (6):
  - UCLA Center for Vaccine Research, Torrance, California
  - Maryland CARES, College Park, Maryland
  - Center for Vaccine Development, St Louis, Missouri
  - Univ of Rochester Medical Center, Rochester, New York
  - Inf Dis Clinic at Gamble Research Clinic and Bethesda Hosp, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas